CLINICAL TRIAL: NCT07284979
Title: A Phase 3, Randomized, Active- and Placebo-Controlled, Partially-Blinded Study to Compare the Efficacy and Safety of KAI-9531 Administered Once Weekly Versus Semaglutide and Placebo in Participants Living With Obesity Who Do Not Have Diabetes
Brief Title: Efficacy and Safety of KAI-9531 Administered Once Weekly Compared With Semaglutide and Placebo in Participants Living With Obesity Who Do Not Have Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kailera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K9531-3107; 2025-523511-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Obesity; KAI-9531; Glucagon-like peptide-1; GLP-1; Semaglutide; Glucose-dependent Insulinotropic Peptide; GIP
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participant and investigator will be blinded for participants randomized to KAI-9531 or placebo until the study is complete. Semaglutide will be provided open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- KAI-9531: Dose 1 (Experimental): Participants will receive Dose 1 of KAI-9531 once weekly.
  Interventions: Drug: KAI-9531
- KAI-9531: Dose 2 (Experimental): Participants will receive Dose 2 of KAI-9531 once weekly.
  Interventions: Drug: KAI-9531
- Semaglutide (Active Comparator): Participants will receive semaglutide once weekly.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive placebo matched to KAI-9531 once weekly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KAI-9531 — SC Injection
  Arms: KAI-9531: Dose 1; KAI-9531: Dose 2
Drug: Semaglutide — SC Injection
  Other Names: Wegovy
  Arms: Semaglutide
Drug: Placebo — SC Injection
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate that KAI-9531 subcutaneous (SC) injection once weekly is superior to semaglutide SC once weekly and to placebo SC once weekly on percent change in body weight.

ELIGIBILITY:
Key Inclusion Criteria:

* BMI ≥35 kilograms per square meter (kg/m^2).
* History of at least 1 self-reported unsuccessful effort to lose weight with diet and exercise within the prior 6 months.

Key Exclusion Criteria:

* Current diagnosis or history of diabetes mellitus.
* Started medications within 3 months prior to Screening that may cause significant weight gain, including, but not limited to, tricyclic antidepressants, atypical antipsychotics, and mood stabilizers.
* Unstable weight defined as self-reported change in body weight exceeding 5% within the 3 months prior to Screening.
* Family or personal history of multiple endocrine neoplasia Type 2 or medullary thyroid cancer.
* Uncontrolled hypertension or unstable cardiovascular disease.
* History of chronic or acute pancreatitis.
* Known clinically significant gastric-emptying abnormality or chronic treatment with medications that directly affect gastrointestinal motility.
* History of suicide attempt.
* History of significant active or unstable Major Depressive Disorder (MDD) or other severe psychiatric disorder.
* Received treatment with semaglutide, tirzepatide, glucagon-like peptide-1 receptor (GLP-1R) agonist, GLP-1/glucose-dependent insulinotropic polypeptide (GIP), or glucagon receptor agonist within 3 months prior to Screening.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-04-17 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Body Weight at Week 76 | Baseline, Week 76

SECONDARY OUTCOMES:
Percentage of Participants with ≥10%, ≥15%, ≥20% and ≥25% Reduction in Body Weight | Baseline, Week 76
Change From Baseline in Waist Circumference | Baseline, Week 76
Change From Baseline in Absolute Body Weight | Baseline, Week 76
Percentage of Participants with ≥5% Reduction in Body Weight | Baseline, Week 76
Change From Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 76
Percent Change From Baseline in Fasting Triglycerides | Baseline, Week 76
Percent Change From Baseline in Fasting High-density Lipoprotein (HDL)-cholesterol | Baseline, Week 76
Percent Change From Baseline in Fasting Non-HDL-cholesterol | Baseline, Week 76
Change From Baseline in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score | Baseline, Week 76
Percentage of Participants with ≥30% Reduction in Body Weight | Baseline, Week 76
Change From Baseline in Body Mass Index (BMI) | Baseline, Week 76
Change From Baseline in Control of Eating Questionnaire (CoEQ) Craving Control Score | Baseline, Week 76
Change From Baseline in CoEQ Positive Mood Score | Baseline, Week 76
Change From Baseline in CoEQ Craving for Sweets Score | Baseline, Week 76
Change From Baseline in CoEQ Craving for Savory Food Score | Baseline, Week 76
Change From Baseline in CoEQ Hunger Score | Baseline, Week 76
Change From Baseline in CoEQ Satiety Score | Baseline, Week 76
Change From Baseline in CoEQ Combined Score | Baseline, Week 76
Change From Baseline in Food Noise Questionnaire (FNQ) Score | Baseline, Week 76
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Week 80
Number of Participants With Anti-drug Antibodies (ADAs) | Up to Week 80
Number of Participants With Neutralizing Antibodies (Nabs) | Up to Week 80
Plasma Concentrations of KAI-9531 | Up to Week 76

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Kailera Clinical Site, Northridge, California
  - Kailera Clinical Site, Stamford, Connecticut
  - Kailera Clinical Site, Albany, Georgia
  - Kailera Clinical Site, Shreveport, Louisiana
  - Kailera Clinical Site, Spartanburg, South Carolina
  - Kailera Clinical Site, Manassas, Virginia
  - Kailera Clinical Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No